CLINICAL TRIAL: NCT01264094
Title: A Study to Evaluate the Efficacy and the Change of sAg Levels in Chronic Hepatitis B Patients Receiving Clevudine Treatment Over the Long Period
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Kwan Sik Lee/Gangnam Severance Hospital, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLV-408
Record Dates: First submitted 2010-12-19; First posted 2010-12-21 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — clevudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clevudine — clevudine 30 mg qd

SUMMARY:
The purpose of this study is to evaluate the efficacy and the Change of sAg Levels in Chronic Hepatitis B Patients Receiving Clevudine Treatment Over the Long Period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years and older.
2. Patient is documented to be HBsAg positive for > 6 months and HBV DNA positive.
3. Patient is HBeAg positive or negative.
4. Patient has ALT levels ≥ 80 IU/L
5. Patient who is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
2. Patients previously treated with interferon within the previous 3 months.
3. Patients previously treated with clevudine, lamivudine, adefovir, entecavir, telbivudine or any other investigational nucleoside for HBV infection.
4. Patient is coinfected with HCV, HDV or HIV.
5. Patient is pregnant or breast-feeding.
6. Patient has a clinically relevant history of abuse of alcohol or drugs.
7. Patient has a significant immunocompromised, gastrointestinal, renal, hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic(except HCC)or allergic disease or medical illness that in the investigator's opinion might interfere with therapy.
8. Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBV DNA below the assay limit of detection

SECONDARY OUTCOMES:
The change of HBV DNA from the baseline.
Proportion of patients with HBeAg loss and/or seroconversion.
Biochemical improvement (e.g. ALT normalization).
Proportion of sAg loss

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea